CLINICAL TRIAL: NCT02855229
Title: Novel Cross-Species Neurophysiological Assays of Reward and Cognitive Domains
Status: Completed | Type: Observational
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Diego Pizzagalli, Director, Center for Stress, Depression and Anxiety Research, Mclean Hospital
Other Study IDs: 2015P001757/MGH
Record Dates: First submitted 2016-07-11; First posted 2016-08-04 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2023-01

CONDITIONS: Translational Electrophysiology
Keywords: Translational; Electrophysiology
MeSH Terms: interventions — Methylphenidate; Modafinil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood samples, saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: No

GROUPS / COHORTS (4):
- Phase 1 Participants [No Study Drug]: Phase 1 participants are not being assigned to any study drug.
- Phase 2 Participants [Placebo]: Phase 2 participants that are randomly assigned to the placebo.
- Phase 2 Participants [Methylphenidate]: Phase 2 participants that are randomly assigned to take methylphenidate.
  Interventions: Drug: Methylphenidate
- Phase 2 Participants [Modafinil]: Phase 2 participants that are randomly assigned to take modafinil.

INTERVENTIONS:
Drug: Methylphenidate — cross-over, single-dose intervention
  Other Names: Modafinil
  Groups: Phase 2 Participants [Methylphenidate]

SUMMARY:
The overarching goal of this multi-disciplinary research program is to develop and optimize new cross-species translational assessments of reward and cognition that will not only be assessed in parallel in humans and rats, but also produce neurophysiological and behavioral metrics that can be objectively compared across species. The research will build on prior studies by further developing and optimizing (in Phase 1), then validating via pharmacological challenge (in Phase 2), the following assays in both humans and rats:

1. advanced neurophysiological and computational modeling techniques to record and analyze EEG activity within and across species; and
2. behavioral assessments of reward learning, cognitive control, and cognitive flexibility will be analyzed within and across species.

The second phase of the study will test the translational validity of these assays, by assessing the impact of a targeted drug on task performance and EEG activity in both species.

DETAILED DESCRIPTION:
The overarching goal of this multi-disciplinary research program is to develop and optimize new translational assessments of reward and cognition that will produce neurophysiological and behavioral metrics that enable objective comparison of drug effects.

Phase 1 (2016-2018) will seek to develop and optimize computer-based tasks to measure of reward learning and cognition, to be administered during an EEG examination. Each participant will be asked to come for a single visit to complete a brief psychological assessment (interview and surveys), then perform two of the computer-based tasks while EEG data are collected. The three tasks are the Flanker Task, the Reversal Learning Task, and the Probabilistic Reward Task (PRT).

In Phase 2 (2018-2021), a new set of participants will be enrolled for four visits. At the first visit they will have a brief psychological assessment (interview and surveys). They will then be assigned to one of the tasks developed during Phase I, and they will also be assigned to one of the study drugs: modafinil (a cognitive enhancer) or methylphenidate (a dopamine enhancer). At the second, third, and fourth visit, the subject will be given their drug in one of the three doses: a low dose, a higher dose, and a placebo. They will then perform the assigned task during an EEG exam.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Right-handed

Exclusion Criteria:

* acute or chronic medical, neurological, or psychiatric illness
* any past/current diagnosis of mental health disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), including alcohol or substance abuse;
* use of any psychotropic medications in the past 6 months
* Current depressed mood (Beck Depression Inventory (BDI-II) score < 6)
* Current use of aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), warfarin, and other anticoagulants
* History of cocaine, stimulant, and other dopaminergic drug use (e.g., amphetamine, methylphenidate)
* Positive toxicology screen at any session

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Feedback-related positivity (FRP) amplitudes over frontocentral scalp regions in response to rewarded trials versus no-reward trials. | 1 Day
  Relative FRP response is the primary outcome measure for the probabilistic reward task (PRT) used in Phase 1.
Event-related negativity (ERN) amplitudes over frontocentral scalp regions in response to correct trials versus incorrect trials. | 1 Day
  Relative ERN response is the primary outcome measure for the flanker task.
Feedback-related negativity (FRN) amplitudes over frontocentral scalp regions in response to negative feedback versus positive feedback. | 1 Day
  Relative FRN response is the primary outcome measure for the reversal learning task.
Behavioral Performance on the Flanker Task | 1 Day
  The Flanker Task is a cognitive task that measures response inhibition to assess the ability to suppress responses that are inappropriate in a particular context.
Behavioral Performance on the Reversal Learning Task | 1 Day
  The task involves learning 'rule' which determine which of two abstract stimuli are selected. The rule changes in the middle of the block, and the goal is to see how quickly the participant can adapt to the rule change. Feedback is probabilistic.

CONTACTS AND LOCATIONS:
Overall Officials: Diego A Pizzagalli, PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared via NIMH Data Archive (as part of data submission agreement)
Time Frame: All collected IPD are shared every 6 months (1/15 and 7/15 of each year). Uploading will begin in 2019.
Access Criteria: Investigators may request for access for approval by the NIMH.